CLINICAL TRIAL: NCT05428241
Title: The Effect of Motivational Interviews on Coping, Functionality, Treatment Adherence and Quality of Life in Patients With Bipolar Disorder
Brief Title: Motivational Interviewing in Patients With Bipolar Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Halis YILMAZ, Principal Investigator-PhD Student, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 60116787-020-155550
Record Dates: First submitted 2022-06-14; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Motivational Interviews; Bipolar Disorder
Keywords: Motivational Interviews; Bipolar Disorder; Coping; Functionality; Treatment Adherence; Quality of Life
MeSH Terms: conditions — Bipolar Disorder; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: Randomized controlled pre-post test design
Who Masked: Participant, Care Provider
Masking Description: Participants and caregivers were not informed about intervention content and measurements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Study group intervention consists 6-session Motivational Interviews and 3-month follow-up.
  Interventions: Behavioral: Assigned Interventions
- No Intervention (No Intervention): Control group receives general care and the training booklet at the end of the study. Also includes 3-month follow-up.

INTERVENTIONS:
Behavioral: Assigned Interventions — Behavioral: 6 sessions of Motivational Interviewing and 3-month follow-up. 6 sessions of Motivational Interview will be applied to the working group. All sessions will be in the form of face-to-face meetings. Each interview will take an average of 45-60 minutes. With this intervention, it was aimed to increase the levels of coping with motivational interviewing, functionality, adherence to treatment and quality of life in bipolar disorder patients. Study data consists of personal information form, Morisky Treatment Adherence Scale (MMAS), World Health Organization Quality of Life Scale, Short Form (WHOQOL-BREF), Assessment of Coping Attitudes Inventory (COPE), Bipolar Disorder Functioning Questionnaire (BDFQ). Data will be analyzed pre-intervention, post-intervention and 3 months post-intervention. A drug and device will not be administered to participants.
  Arms: Experimental

SUMMARY:
Introduction: A poor therapeutic relationship, poor quality of life, impaired functioning, ineffective coping methods, and lack of motivation It is associated with poor adjustment (to symptoms, treatment, and environment) in patients with bipolar disorder. In order to achieve better compliance and results, the therapeutic relationship, coping skills, quality of life and functionality should be improved by increasing the motivation of individuals.

Purpose: This study was planned to examine the effects of motivational interviewing on coping, functioning, adherence to treatment and quality of life in patients with bipolar disorder.

Methods: In this single-blind, randomized controlled trial, simple randomization method and pretest-posttest control group design, experimental research design will be used. The work will take place at: Pamukkale University Health Research and Application Center, Psychiatric Hospital from July 2021 to February 2022 and including 48 individuals (24 in the experimental group and 24 in the control group). Working data it will be collected using personal information form, Morisky Medication Adherence Scale (MMAS), The World Health Organization Quality of Life Scale, the Short Form (WHOQOL-BREF), Assessment of Coping Attitudes Inventory (COPE), and Bipolar Disorder Functioning Questionnaire (BDFQ). The researchers will conduct a 6- session of motivational interviewing with the participants in the experimental group. No intervention will be made in the control group. Data will be analyzed on a pre-intervention, post-intervention and post-intervention 3 months (follow-up) basis.

DETAILED DESCRIPTION:
Bipolar disorder is a serious mental disorder with depressive, manic or hypomanic episodes, which is completely normal or thought to be associated with minimal symptom levels, and is known to cause high mortality, morbidity, and loss of function in almost all areas. Gaining functionality in patients with bipolar disorder, improving their compliance with treatment and quality of life, and helping them to cope with stress are among the most important goals of treatment.

In individuals with bipolar disorder, stressful life events can lead to early onset of the disease, more frequent depression, psychotic symptoms, and problems such as anxiety. It is stated that patients with bipolar disorder have problems in interpersonal relationships and problems in coping with stress. When patients with a diagnosis of bipolar disorder in remission encounter a stressful life event, their functionality in the areas of work/school, family, and friends may be affected or even impaired.

Since bipolar disorder is a chronic disease, it is stated that it affects people's lives in terms of their functionality during remission periods as well as during attacks. Marriage-related problems, economic difficulties and substance use, together with the risk of suicide and irregular work history, can cause dysfunction in patients in wide psychosocial areas. It has been reported that the quality of life of patients whose functionality is impaired during the remission period also deteriorates.

Due to the early onset of bipolar disorder, the length of time until diagnosis, and inadequate treatment, it harms patients in terms of quality of life and expected psychosocial development. It is stated that depressive symptoms, being a woman, the length of time until the diagnosis, low socioeconomic and educational level are factors that increase the deterioration in the quality of life in rural areas in patients with bipolar disorder. In addition, the presence of another comorbidity accompanying bipolar disorder (anxiety, alcohol-substance addiction, etc.) also affects the quality of life. However, when the clinical studies on the disorder are examined, it is seen that the lack of compliance of the patients with the treatment causes the quality of life to deteriorate.

In bipolar disorder, low treatment compliance is caused by the patient's insufficient insight into the disease, reservations about the drug, negative clinical course of the disease, insufficient social and environmental support, economic difficulties, insufficient information about treatment, unfavorable conditions of the living environment or treatment center, the patient's and his/her environment's drug addiction. treatment and attitude towards bipolar disorder, prejudices caused by drug use in society, and cultural beliefs.

Poor therapeutic relationship, poor quality of life, impaired functioning, ineffective coping methods, and lack of motivation It is associated with poor adjustment (to symptoms, treatment, and environment) in patients with bipolar disorder. In order to achieve better compliance and results, the therapeutic relationship, coping skills, quality of life and functionality should be improved by increasing the motivation of individuals. Nurses need to establish a therapeutic relationship in order for the nursing care to produce effective results during the recovery process of these patients.

In this study, it is thought that Motivational Interviewing may be effective in increasing effective coping skills, functionality, adherence to treatment and quality of life in patients with bipolar disorder, and may shed light and guide psychiatric nursing interventions.

ELIGIBILITY:
Inclusion Criteria:

* To be at least primary school graduate,
* Be willing to participate in research.
* Being between the ages of 18-65,
* Able to understand and speak Turkish,
* Patients who can understand scales and forms,
* Being registered in the euthymic period and Denizli Pamukkale University Health Research and Application Center Psychiatry Department Community Mental Health Center unit
* To have a diagnosis of bipolar disorder I-II for at least 1 year according to DSM-5 (The Diagnostic and Statistical Manual of Mental Disorders) diagnostic criteria.

Exclusion Criteria:

* Being under the age of 18 and over the age of 65,
* Being illiterate in Turkish,
* Having Mental Retardation,
* Being diagnosed with a mental illness other than bipolar disorder according to the DSM-5 (The Diagnostic and Statistical Manual of Mental Disorders) diagnostic criteria,
* Being in an manic or depressed attack period,
* Patients who have received or are continuing a similar education program.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
Morisky Treatment Adherence Scale | Change from baseline Morisky Treatment Adherence Scale at 3 months
  The scale consists of four likert-type two-answer questions. The questions are in the form of closed-ended "yes and no". If all questions are answered "no", drug compliance is considered high, if "yes" is answered for one or two questions, drug compliance is considered medium, if yes to three or four questions, drug compliance is considered low. In the scale, 0-1 points indicate low, 2-3 points moderate, and 4 points high adherence to treatment.
The World Health Organization Quality of Life Instrument, Short Form | Change from baseline The World Health Organization Quality of Life Instrument, Short Form at 3 months
  It is a scale developed from the World Health Organization's WHOQOL-100 to assess quality of life. WHOQOL-BREF consists of 26 questions and four areas selected from WHOQOL-100. These 4 areas are physical, mental, social relations and environmental areas. The 3rd, 4th and 26th items of the scale are reverse scored. WHOQOL-BREF has Likert-type scoring ranging from 1 to 5. As the score obtained from the sub-domains of the scale increases, the quality of life increases.
Assessment of Coping Attitudes Inventory | Change from baseline Assessment of Coping Attitudes Inventory at 3 months
  There are 60 questions in total and 15 subscales, each consisting of four questions. Each subscale is answered over four options. These answers are: 1=I would never do anything like this; 2=I do very little like this; 3=I do this moderately; 4=I usually do it like this. Positive reinterpretation and growth, use of beneficial social support, active coping, religious coping, joking, holding back, use of emotional social support, acceptance, suppression of other occupations, and planning subscales represent adaptive coping methods, while mental distancing, problem-focused and problem-focused and expressing emotions, denial, behavioral distancing, and substance use subscales are considered as maladaptive coping methods. As a result, the high scores to be obtained from the subscales give the possibility to comment on which coping attitude is used more by the individual.
Bipolar Disorder Functioning Questionnaire | Change from baseline Assessment of Coping Attitudes Inventory at 3 months
  The scale is in triple Likert type and the items are calculated by giving 1 point 'no or nothing', 2 points 'partly or sometimes', and 3 points 'yes or always'. The 1st and 3rd questions in the emotional functionality subscale, the 5th and 7th questions in the mental functionality subscale, the 8th, 10th and 11th questions in the sexual functionality subscale, and the 49th, 50th and 51st questions in the work subscale are reversed. is scored. The total score can range from 52 to 156. The scale does not have a cutoff score, and as the score increases, functionality also increases.

SECONDARY OUTCOMES:
Number of health care uses | Change in the number of initial health care use in the 3rd month
  According to the patient's declaration, number of hospitalizations.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Yiğitoğlu, PhD, Study Director — Pamukkale University; Halis Yılmaz, Msc, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Faculty of Health Science, Departmant of Psychiatric Nursing, Denizli, Denizli, Kınıklı Kampus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study results will be announced in a publication
Supporting Information: Study Protocol, SAP
Time Frame: Findings can be shared after the study has been published.
Access Criteria: The sociodemographic and disease-related characteristics of the participants, the pre-post-test and follow-up findings including the answers to the research questions and statistical analyzes will be shared.

REFERENCES:
- [Result] Pakpour AH, Modabbernia A, Lin CY, Saffari M, Ahmadzad Asl M, Webb TL. Promoting medication adherence among patients with bipolar disorder: a multicenter randomized controlled trial of a multifaceted intervention. Psychol Med. 2017 Oct;47(14):2528-2539. doi: 10.1017/S003329171700109X. Epub 2017 Apr 27. PMID 28446253
- [Result] McKenzie K, Chang YP. The effect of nurse-led motivational interviewing on medication adherence in patients with bipolar disorder. Perspect Psychiatr Care. 2015 Jan;51(1):36-44. doi: 10.1111/ppc.12060. Epub 2014 Jan 17. PMID 24433493
- [Result] Laakso LJ. Motivational interviewing: addressing ambivalence to improve medication adherence in patients with bipolar disorder. Issues Ment Health Nurs. 2012 Jan;33(1):8-14. doi: 10.3109/01612840.2011.618238. PMID 22224961
- [Result] Ertem MY, Duman ZC. The effect of motivational interviews on treatment adherence and insight levels of patients with schizophrenia: A randomized controlled study. Perspect Psychiatr Care. 2019 Jan;55(1):75-86. doi: 10.1111/ppc.12301. Epub 2018 Jun 11. PMID 29888541
- [Result] Goldstein TR, Krantz ML, Fersch-Podrat RK, Hotkowski NJ, Merranko J, Sobel L, Axelson D, Birmaher B, Douaihy A. A brief motivational intervention for enhancing medication adherence for adolescents with bipolar disorder: A pilot randomized trial. J Affect Disord. 2020 Mar 15;265:1-9. doi: 10.1016/j.jad.2020.01.015. Epub 2020 Jan 7. PMID 31957686